CLINICAL TRIAL: NCT00533715
Title: Forced Inspiratory Flow Volume Curve in Healthy Young Children
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-03-2303-BA-CTIL
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Healthy
Keywords: Inspiratory Spirometry; Preschool Children; Computer games; Health

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- >100: The study included healthy children (2.5-6.5 years old) from a number of public kindergartens. An initial screening questionnaire based on the ATA-DLD-78-A for adults, adapted for children and translated into Hebrew, concerning the child's birth, past and present health status, was completed by the parents.
  Exclusion criteria: Previous symptoms or treatment for asthma, current respiratory symptoms or other present respiratory diseases.

SUMMARY:
Spirometry testing should include both expiratory and inspiratory measurements as it may influence the expiratory flow volume curve indices. The ability to inhale medication may by judged by inspiratory flows. However, the inspiratory portion of the forced flow/volume maneuver in young healthy children has not yet been described.Objectives: To document and analyze the forced inspiratory flow volume curve indices in healthy young children.

Settings: Community kindergartens around Israel. participants; Healthy preschool children (age 2.5-6.5 years).

Methods: The teaching method included multi-target, interactive spirometry games (SpiroGame®) and accessory games for inspiration (e.g. inspiratory whistle).

Results: One hundred and fourteen of 157 children performed duplicate full adequate inspiratory maneuvers. Repeatability between two maneuvers was 5.6%, 4.0%, 5.1%, 7.3% for inspiratory capacity (IVC), forced inspiratory capacity (FIVC), peak inspiratory capacity (PIF), and mid inspiratory flow (MIF50), respectively. Inspiratory flow indices were significantly lower than the parallel expiratory flow indices and the time to reach PIF was significantly slower than the time to reach peak expiratory flow (meanSD; 22921ms vs. 92 8ms; p<0.0001). The shape of the inspiratory curve was parabolic and did not change with age. Predicted equations that were formed were in agreement with the extrapolated prediction equation values of older children.

We found that the majority of healthy young children can produce reliable inspiratory curves. Our results provide a framework for reference equations for inspiratory flow volume curve in the young ages. The clinical applications of these equations are yet to be explored.

DETAILED DESCRIPTION:
Study protocol: The study included healthy children (according to questionnaire) in their early childhood. Any children with previous symptoms or present treatment for asthma, respiratory symptoms (cough, post nasal drip, pneumonia, rhinitis) other respiratory diseases were excluded from the study. Forced maneuvers were measured with a commercial spirometer, ZAN100 (ZAN Messgerate, Oberthulba, Germany). The spirometer software included online analysis of inspiratory and expiratory maneuvers. The curves were monitored on the computer screen to ensure best effort. The software also included an incentive-guided spirometry game. Inspiratory indices were not part of the games, therefore efforts were continued until the child could not pass the former inspiratory attempt any further. Healthy children performed the tests in a designated room in the kindergarten. Tests were performed in a standing position without a nose-clip. Maneuvers were repeated to obtain best possible efforts on at least three technically acceptable maneuvers. Technically acceptable curves were stored and the three consecutive curves with the maximal inspiratory maneuvers were analyzed for the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy children between 3-6 years old

Exclusion Criteria:

* Past or present respiratory lung disease

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2003-01; Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barak Asher, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- The Edmond and Lily Safra Children's Hospital, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- See also: Vilozni D, et al. The role of computer games in measuring spirometry in healthy and "asthmatic" preschool children. Chest. 2005 Sep;128(3):1146-55. — http://www.ncbi.nlm.nih.gov/sites/entrez